CLINICAL TRIAL: NCT02112656
Title: A Phase III, Randomized, Double Blind, Dummy-Controlled Study of ThermoDox® (Lyso-Thermosensitive Liposomal Doxorubicin-LTLD) in Hepatocellular Carcinoma (HCC) Using Standardized Radiofrequency Ablation (RFA) Treatment Time ≥ 45 Minutes for Solitary Lesions ≥ 3 cm to ≤ 7 cm
Brief Title: Study of ThermoDox With Standardized Radiofrequency Ablation (RFA) for Treatment of Hepatocellular Carcinoma (HCC)
Acronym: OPTIMA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Imunon (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 104-13-302
Record Dates: First submitted 2014-04-10; First posted 2014-04-14 (Estimated); Results first posted 2024-08-20 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-07

CONDITIONS: Hepatocellular Carcinoma
Keywords: Carcinoma; Carcinoma, Hepatocellular; Neoplasms, Glandular and Epithelial; Neoplasms by Histologic Type; Neoplasms; Adenocarcinoma; Liver Neoplasms; Digestive System Neoplasms; Neoplasms by Site; Digestive System Diseases; Liver Diseases; Doxorubicin; Antibiotics, Antineoplastic; Antineoplastic Agents; Therapeutic Uses; Pharmacologic Actions
MeSH Terms: conditions — Carcinoma, Hepatocellular; Carcinoma; Neoplasms, Glandular and Epithelial; Neoplasms by Histologic Type; Neoplasms; Adenocarcinoma; Liver Neoplasms; Digestive System Neoplasms; Neoplasms by Site; Digestive System Diseases; Liver Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ThermoDox 50 mg/m2 (Experimental): ThermoDox plus standardized RFA using standardized treatment dwell time for solitary HCC lesions ≥ 3.0 cm to ≤ 7.0 cm
  Interventions: Drug: ThermoDox
- Dummy infusion (Placebo Comparator): standardized RFA alone using standardized treatment dwell time for solitary HCC lesions ≥ 3.0 cm to ≤ 7.0 cm
  Interventions: Drug: Dummy infusion

INTERVENTIONS:
Drug: ThermoDox — Thermally Sensitive Liposomal Doxorubicin 50 mg/m2 Single 30 minute intravenous infusion
  Other Names: Lyso-Thermosensitive Liposomal Doxorubicin (LTLD)
  Arms: ThermoDox 50 mg/m2
Drug: Dummy infusion — Sodium Chloride 0.9% or 5% Dextrose (D5W), Single 30 minute intravenous infusion
  Other Names: Placebo
  Arms: Dummy infusion

SUMMARY:
The purpose of this study is to determine whether ThermoDox, a thermally sensitive liposomal doxorubicin, is effective in the treatment of non-resectable hepatocellular carcinoma when used in conjunction with standardized radiofrequency ablation (sRFA).

DETAILED DESCRIPTION:
This is a Phase III, randomized, double blind, dummy controlled safety and efficacy study of ThermoDox plus sRFA compared to sRFA plus dummy infusion using standardized treatment dwell time for solitary HCC lesions ≥ 3.0 cm to ≤ 7.0 cm. An sRFA treatment for this protocol is defined as the dwell time of ≥ 45 minutes measured from the first activation of the RFA probe through removal of the RFA probe after the final ablation cycle or deployment.

The 50 mg/m2 ThermoDox or dummy infusion will be administered IV over 30 minutes. As part of blinded pre-medication ThermoDox treated subjects will receive 20 mg of dexamethasone orally 24 hours prior to the drug infusion for infusion reaction prophylaxis. Subjects on the control arm will receive a matching dummy pre-medication pill orally at 24 hours prior to infusion of the study treatment. Thirty minutes prior to receiving the ThermoDox infusion, subjects will receive a blinded dose of 20 mg of IV dexamethasone, 50 mg IV diphenhydramine and either 50 mg of IV ranitidine or 20 mg of IV famotidine. Subjects on the control arm will receive a masked dummy pre-medication pill orally at 24 hours prior to infusion of the study medication, and a dummy infusion 30 minutes prior to dummy infusion of Sodium Chloride 0.9% or 5% Dextrose (D5W). RFA will be initiated approximately at a minimum of 15 minutes after the initiation of study drug infusion and should be completed no later than 3 hours after study drug infusion initiation. The goal is to reach a > 45 minute dwell time which can be achieved by employing at least four ablation cycles or deployments in order to ablate the tumor as well as a 360º 1.0 cm tumor-free margin surrounding the tumor.with an estimated overall procedure time of less than 3 hours.

A subject who has an incomplete ablation is eligible for 1 retreatment procedure within 21 days after the radiological imaging exam showing residual disease at Day 28. Subjects will be retreated only once with the same RFA equipment and treatment assigned at randomization. Subjects with a complete ablation after retreatment will be followed both for PFS and for OS.

If after 2 ablations the subject has local, distant intrahepatic, or extrahepatic HCC, then the subject will be considered a treatment failure and will have met the PFS endpoint. The subject will be followed for OS every 3 months. Among subjects who are not treatment failures, five repeat treatments are permitted to treat a recurrent lesion or to treat newly-identified local or distant intrahepatic lesions at the Investigator's discretion after the PFS endpoint is reported and with agreement from the Sponsor. The subject must be eligible for retreatment consistent with the safety eligibility criteria and will be retreated with the same randomized treatment.

CT or MRI imaging will be used to assess the effectiveness of the ablation therapy. The blind will be maintained at the level of the imaging reads. Investigator determined radiological progression must be observed and recorded prior to beginning alternate treatments for HCC. Posttreatment imaging will be obtained at months 1, 5, 9, 13, 17, 21, 25, then every 6 months (+/- 2 weeks) until radiological progression is seen. Adverse event assessments and laboratory examinations will occur at each visit. All subjects will be monitored throughout the investigational period.

Patients that meet inclusion/exclusion criteria may be at risk for contrast-induced nephropathy (CIN) when undergoing the required CT with contrast procedures. The investigators must be mindful of the risk factors associated with CIN and employ strategies to reduce the risk of CIN. In subjects with diabetes or borderline renal function (creatinine greater than 1.5 mg/dL) special precautions (e.g. hydration, contrast dose reduction, follow up creatinine determination) should be employed. An accepted procedure is adequate intravenous volume expansion with isotonic saline (1.0 - 1.5 mL/kg per hour) for 3-12 hours before the procedure and continued for 6-24 hours if clinically indicated and based on the treating physician's medical judgment.

All randomized subjects will be followed for safety and overall survival.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥ 18 years of age.
2. Diagnosed with a single HCC lesion ≥ 3.0 cm but ≤ 7.0 cm in maximum diameter based on diagnosis at screening.

   * Subjects meeting the American Association for the Study of Liver Disease (AASLD) criteria may be randomized without a biopsy, but will undergo a biopsy during the RFA procedure unless contraindicated or unattainable.
   * Subjects not meeting the AASLD criteria for HCC will need a biopsy to confirm HCC prior to randomization.
3. Be an appropriate candidate for receiving RFA as a medically indicated treatment as evaluated by the following factors:

   * The position and accessibility of the target lesion allows for the safe administration of multiple ablation cycles or deployments to achieve a probe dwell time of ≥ 45 minutes.
   * Not a candidate for surgical resection according to the local guidelines for resection and in the Investigator's judgment.
4. Child-Pugh Class A without either current encephalopathy or ascites.
5. Left Ventricular Ejection Fraction (LVEF) ≥ 50%.
6. Eastern Cooperative Oncology Group (ECOG) performance status 0.
7. Willing to sign an informed consent form, indicating awareness of the investigational nature of this study that is in keeping with the policies of the institution.

Exclusion Criteria:

1. Is scheduled for liver transplantation
2. Expected ablation volume > 30% of total liver volume or removal of 3 hepatic segments
3. More than 1 lesion identified during baseline.
4. Have previously received therapeutic treatment for HCC outside the study protocol or is expected to receive concomitant HCC treatment prior to PFS event.
5. Have serious medical illnesses including, but not limited to, congestive heart failure, myocardial infarction or cerebral vascular accident within the last six months, or life threatening cardiac arrhythmias.
6. Have previously received any anthracycline outside the protocol
7. Have extrahepatic metastasis.
8. Have portal or hepatic vein tumor invasion/thrombosis.
9. Have body temperature >101ºF (38.3ºC) immediately prior to study treatment.
10. Baseline laboratories (repeat lab tests are permitted to evaluate eligibility during the Screening Period. Lab results must be within protocol range prior to study treatment.)

    * Absolute neutrophil count < 1500/mm3
    * Platelet count < 75,000/mm3
    * Hgb < 10.0 g/dL (unless the hemoglobin value has been stable, the subject is cardiovascularly stable, asymptomatic and judged able to withstand the RFA procedure) Note: If clinically indicated, subjects may receive platelets or packed red blood cell (RBC) transfusions and be re-evaluated after condition is treated.
11. Baseline Chemistry

    * Serum creatinine ≥ 2.5 mg/dL or calculated creatinine clearance (CrCl) ≤25.0 mL/min.
    * Serum bilirubin > 3.0 mg/dL.
    * Serum albumin < 2.8 g/dL.
12. Have any known allergic reactions to any of the drugs or liposomal components or intravenous imaging agents that prohibit the ability to complete the imaging requirements.
13. Are pregnant or breast-feeding. In women of childbearing potential, a negative serum pregnancy test is required prior to study treatment.
14. Women of childbearing potential and men who are not practicing an acceptable form of birth control (i.e. diaphragm, cervical cap, condom, surgical sterility or birth control pills. Women whose partner has or men who have undergone a vasectomy must use a second form of birth control).
15. Have INR > 1.5 times the institution's upper normal limit (UNL), except in subjects who are therapeutically anticoagulated for medical conditions unrelated to HCC such as atrial fibrillation. Subjects may be re-screened after condition is treated or anticoagulant is withheld.
16. Have contraindications to receiving doxorubicin hydrochloride (HCl).
17. Are being treated with other investigational agents.
18. Use of an investigational drug outside this study within 30 days or 5 half-lives, whichever is longer, preceding the first dose of study medication.
19. Have other concurrent malignancy (subjects with treated squamous cell carcinoma of the skin or basal cell carcinoma of the skin may be included), evidence of extrahepatic cancer from their primary malignancy, or ongoing, medically significant active infection.
20. HIV positive.
21. NYHA class III or IV functional classification for heart failure.
22. Evidence of hemachromatosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 554 (Actual)
Dates: Start 2014-06; Primary Completion 2020-04-27 (Actual); Study Completion 2020-04-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo Lencioni, MD, Study Chair — University of Pisa; Ronnie Tung Ping Poon, MD, Study Chair — Hong Kong University; Chen Min Hua, MD, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (61):
- UCLA Department of Medicine, Los Angeles, California, United States
- Toronto General Hospital, Toronto, Ontario, Canada
- China (17):
  - Mengchao Hepatobiliary Hospital of Fujian Medicatl University, Fuzhou, Fujian
  - Xijing Hospital, Xi'an, Shaanxi
  - Peking University First Hospital, Beijing
  - Beijing Cancer Hospital, School of Oncology, Peking, Beijing
  - 302 Military Hospital of China, Beijing
  - Beijing Hospital of the Ministry of Health, Beijing
  - Chinese PLA General Hospital, Beijing
  - West China Hospital of Sichuan University, Chengdu
  - The Second Hospital of Dalian Medical University, Dalian
  - Guangdong General Hospital, Guangdong
  - Hunan Cancer Hospital, Hunan
  - The First Hospital of Jilin University, Jilin
  - Zhongshan Hospital, Fudan University, Shanghai
  - The Sixth People's Hospital of Shenyang, Shenyang
  - The 3rd Hospital of Tianjing, Tianjin
  - The First Hospital of Zhejiang, Zhejiang
  - Zhejiang Cancer Hospital, Zhejiang
- Germany (4):
  - Institut für Diagnostische und Radiologische Therapie del Uniklinik Frankfurt, Frankfurt
  - Universitaetsklinikum des Saarlandes, Klik fuer Allgemeine Chirurgie, Viszeral-, Gefaess und Kinderchirurgie, Homburg
  - Klinikum rechts der Isar, II. Medizinische Klinik und Poliklinik (Gastroenterologie), München
  - Universitätsklinikum Regensburg, Institut für Röntgendiagnostik, Regensburg
- Queen Mary Hospital, Hong Kong, Hong Kong
- Italy (2):
  - Cisanello Hospital, Division of Diagnostic Imaging and Intervention, Pisa
  - Department of Radiological Sciences and Bioimaging Catholic University of Rome, "A. Gemelli" Hospital, Rome
- University Malaya Medical Centre, Kuala Lumpur, Malaysia
- Philippines (3):
  - Chinese General Hospital and Medical Center, Manila
  - St. Lukes Medical Center, Quezon City
  - Cardinal Santos Medical Center, San Juan City
- Singapore General Hospital, Singapore, Singapore
- South Korea (8):
  - Pusan National University Hospital, Busan
  - Kyungpook National University Hospital, Daegu
  - Kyungpook National University Medical Center, Daegu
  - Inha University Hospital, Incheon
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea, Seoul St.Mary's Hospital, Seoul
- Spain (2):
  - Hospital Madrid Norte Sanchinarro, Madrid
  - Hospital Universitario Marqués de Valdecilla, Santander
- Taiwan (7):
  - Chang Gung Memorial Hospital - Kaohsiung, Kaohsiung City
  - Taipei Medical University-Shuang Ho Hospital, New Taipei City
  - Taichung Veteran General Hospital, Taichung
  - National Cheng Kung University (NCKU) Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Chang Gung Memorial Hospital - Linkou, Taoyuan District
  - National Taiwan University Hospital, Yun-Lin Branch, Yuanlin
- Thailand (5):
  - Siriraj Hospital, Bangkok
  - Maharaj Nakorn Chiang Mai Hospital, Chiang Mai
  - Srinagarind Hospital, Khon Kaen
  - Thammasat University Hospital, Pathum Thani
  - Songklanagarind Hospital, Songkhla
- Vietnam (8):
  - Bach Mai Hospital, Hà Nội, Dong Da District
  - 108 Military Central Hospital, Hà Nội, Hai Ba Trung District
  - Hue Central Hospital, Huế, Vin Ninh Ward
  - Bach Mai Hospital (Hepato-gastroenterology Department), Hanoi
  - Can Tho Oncology Hospital, Hanoi
  - National Cancer Hospital, Hanoi
  - Viet Duc University Hospital, Hanoi
  - People's Hospital 115, Ho Chi Minh City

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ThermoDox 50 mg/m2 | Dummy Infusion
Started | 277 | 277
Completed | 187 | 178
Not Completed | 90 | 99
Not completed — Death | 78 | 82
Not completed — Withdrawal by Subject | 9 | 11
Not completed — Lost to Follow-up | 2 | 4
Not completed — Noncompliance | 1 | 2

BASELINE CHARACTERISTICS:
Population: Baseline participants represent the intent-to-treat (ITT) population.
Groups:
- Total: Total of all reporting groups
Arm/Group | ThermoDox 50 mg/m2 | Dummy Infusion | Total
Number analyzed (Participants) | 277 | 277 | 554
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 62 [28 to 86] | 62 [36 to 90] | 62 [28 to 90]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 65 | 119
  Male | 223 | 212 | 435
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 265 | 257 | 522
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 12 | 19 | 31
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: Overall survival is defined as the time (in months) from the date of randomization to the death from any cause or the end of the study.
Time Frame: All subjects to be contacted every 3 months after radiological progression for vital status reporting. Subjects were followed for OS up to 68 months from randomization.
Population: Intent-to-treat (ITT) population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | ThermoDox 50 mg/m2 | Dummy Infusion
Number analyzed (Participants) | 277 | 277
Months | 58.06 [45.53 to NA] — Not estimable (NA) due to insufficient number of participants reached the event at time of final analysis. | NA [47.93 to NA] — Not estimable (NA) due to insufficient number of participants reached the event at time of final analysis.

2. Secondary Outcome: Progression-free Survival (PFS)
Description: The protocol incorporates modified RECIST developed for HCC clinical research as a basis to evaluate tumor response. PFS here is defined as the time (in months) from the date of randomization to the first date on which one of the following occurs (as determined by CT or MRI scan):
  * Death of any cause
  * Treatment failure (inability to achieve CR after two RFA ± ThermoDox treatment sessions)
  * Progression due to local tumor recurrence after initial CR
  * Progression due to distant intrahepatic tumor recurrence
  * Progression due to extrahepatic tumor recurrence
Time Frame: CT or MRI scan (Chest, Abdomen, Pelvis) done at Baseline and Day 28. Additional imaging done at months 5, 9, 13, 17, 21, 25, then every 6 months until disease progression is seen. Study subjects were followed up to 63 months after randomization.
Population: Intent-to-treat (ITT) population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | ThermoDox 50 mg/m2 | Dummy Infusion
Number analyzed (Participants) | 277 | 277
Months | 19.31 [15.72 to 25.20] | 16.78 [12.86 to 21.32]

ADVERSE EVENTS:
Time Frame: Assess adverse events (AEs) through Day 28 following study treatment. AEs after Day 28 evaluated as possibly, probably or definitely related to the study treatment or the RFA procedure were recorded at any point during the trial and are to be followed until resolution or the patient is clinically stable. In general, all subjects were followed up to 68 months for AE's.
Description: Serious and Other (Not Including Serious) Adverse Events monitored/assessed for the safety-evaluable population and All-Cause Mortality monitored/assessed represent participants who received study treatment.
Arm/Group | ThermoDox 50 mg/m2 | Dummy Infusion
All-Cause Mortality (participants affected / at risk) | 78/277 | 82/277
Serious Adverse Events (participants affected / at risk) | 73/274 | 33/273
Other Adverse Events (participants affected / at risk) | 265/274 | 216/273
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ThermoDox 50 mg/m2 (N=274) | Dummy Infusion (N=273)
Oedema Peripheral (General disorders) | 1 | 0
Multi-Organ Failure (General disorders) | 0 | 1
Portal Vein Thrombosis (Hepatobiliary disorders) | 2 | 1
Cholecystitis Acute (Hepatobiliary disorders) | 1 | 1
Hepatic Failure (Hepatobiliary disorders) | 1 | 0
Hepatic Infarction (Hepatobiliary disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Hepatic Cirrhosis (Hepatobiliary disorders) | 0 | 1
Hepatic Function Abnormal (Hepatobiliary disorders) | 0 | 1
Ischaemic Hepatitis (Hepatobiliary disorders) | 0 | 1
Acute Myocardial Infarction (Cardiac disorders) | 2 | 0
Tachycardia (Cardiac disorders) | 1 | 0
Atrial Fibrillation (Cardiac disorders) | 0 | 1
Atrioventricular Block Complete (Cardiac disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 1 | 0
Procedural Intestinal Perforation (Injury, poisoning and procedural complications) | 1 | 0
Procedural Pain (Injury, poisoning and procedural complications) | 1 | 0
Brachial Plexus Injury (Injury, poisoning and procedural complications) | 0 | 1
Post Procedural Complication (Injury, poisoning and procedural complications) | 0 | 1
Post Procedural Discharge (Injury, poisoning and procedural complications) | 0 | 1
Post Procedural Haematoma (Injury, poisoning and procedural complications) | 0 | 1
Post Procedural Inflammation (Injury, poisoning and procedural complications) | 0 | 1
Cerebrovascular Accident (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Hepatic Encephalopathy (Nervous system disorders) | 1 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary Haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 4
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Drug Hypersensitivity (Immune system disorders) | 1 | 0
Immunosuppression (Immune system disorders) | 1 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Adrenocortical Insufficiency Acute (Endocrine disorders) | 1 | 0
Non-Small Cell Lung Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour Haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Urinary Retention (Renal and urinary disorders) | 1 | 0
Renal Failure Acute (Renal and urinary disorders) | 0 | 1
Renal Impairment (Renal and urinary disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1
Phlebitis (Vascular disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 21 | 1
Febrile Neutropenia (Blood and lymphatic system disorders) | 11 | 0
Bone Marrow (Blood and lymphatic system disorders) | 2 | 0
Leukopenia (Blood and lymphatic system disorders) | 2 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 0
Pneumonia (Infections and infestations) | 4 | 3
Herpes Zoster (Infections and infestations) | 2 | 0
Liver Abscess (Infections and infestations) | 2 | 2
Sepsis (Infections and infestations) | 2 | 2
Urinary Tract Infection (Infections and infestations) | 2 | 0
Diarrhoea Infectious (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0
Neutropenic Sepsis (Infections and infestations) | 1 | 0
Pulmonary Tuberculosis (Infections and infestations) | 1 | 0
Septic Shock (Infections and infestations) | 1 | 1
Subcutaneous Abscess (Infections and infestations) | 1 | 0
Urosepsis (Infections and infestations) | 1 | 0
Wound Infection (Infections and infestations) | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 2 | 1
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 2 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 1 | 0
Apthous Stomatitis (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Intra-Abdominal Haemorrhage (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Duodenal Perforation (Gastrointestinal disorders) | 0 | 1
Haematemesis (Gastrointestinal disorders) | 0 | 1
Lower Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 1
Neutrophil Count Decreased (Investigations) | 4 | 0
White Blood Cell Count Decreased (Investigations) | 3 | 0
Alanine Aminotransferase Increased (Investigations) | 0 | 2
Aspartate Aminotransferase Increased (Investigations) | 0 | 2
Blood Creatinine Increased (Investigations) | 0 | 1
Lymphocyte Count Decreased (Investigations) | 0 | 1
Pyrexia (General disorders) | 2 | 6
Fatigue (General disorders) | 1 | 0
Impaired Healing (General disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ThermoDox 50 mg/m2 (N=274) | Dummy Infusion (N=273)
Neutropenia (Blood and lymphatic system disorders) | 136 | 5
Leukopenia (Blood and lymphatic system disorders) | 28 | 4
Febrile Neutropenia (Blood and lymphatic system disorders) | 12 | 0
Anaemia (Blood and lymphatic system disorders) | 9 | 5
Leukocytosis (Blood and lymphatic system disorders) | 8 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 6 | 5
Bone Marrow Failure (Blood and lymphatic system disorders) | 3 | 0
Pancytopenia (Blood and lymphatic system disorders) | 3 | 0
Lymphopenia (Blood and lymphatic system disorders) | 2 | 0
Disseminated Intravascular Coagulation (Blood and lymphatic system disorders) | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 142 | 1
Rash Erythematous (Skin and subcutaneous tissue disorders) | 2 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 2 | 0
Decubitus Ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 1
Madarosis (Skin and subcutaneous tissue disorders) | 1 | 0
Nail Discolouration (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 1 | 0
Skin Exfoliation (Skin and subcutaneous tissue disorders) | 1 | 0
Skin Reaction (Skin and subcutaneous tissue disorders) | 1 | 0
Subacute Cutaneous Lupus Erythematosus (Skin and subcutaneous tissue disorders) | 1 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis Allergic (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis Atopic (Skin and subcutaneous tissue disorders) | 0 | 1
Skin Ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Neutrophil Count Decreased (Investigations) | 73 | 4
White Blood Cell Count Decreased (Investigations) | 66 | 3
Alanine Aminotransferase Increased (Investigations) | 36 | 45
Aspartate Aminotransferase Increased (Investigations) | 35 | 58
Platelet Count Decreased (Investigations) | 19 | 4
Blood Bilirubin Increased (Investigations) | 11 | 7
Neutrophil Count Increased (Investigations) | 8 | 2
Neutrophil Percentage Decreased (Investigations) | 8 | 0
Haemoglobin Decreased (Investigations) | 7 | 0
Monocyte Percentage Increased (Investigations) | 7 | 0
White Blood Cell Count Increased (Investigations) | 7 | 2
Bilirubin Conjugated Increased (Investigations) | 6 | 3
Blood Pressure Increased (Investigations) | 6 | 7
Lymphocyte Count Decreased (Investigations) | 6 | 2
Lymphocyte Percentage Increased (Investigations) | 6 | 0
Mitochondrial Aspartate Aminotransferase Increased (Investigations) | 6 | 8
Neutrophil Percentage Increased (Investigations) | 6 | 2
Haematocrit Decreased (Investigations) | 5 | 0
Hepatic Enzyme Increased (Investigations) | 5 | 8
Red Blood Cell Count Decreased (Investigations) | 5 | 0
Gamma-Glutamyltransferase Increased (Investigations) | 4 | 1
Blood Albumin Decreased (Investigations) | 3 | 1
Blood Bilirubin Unconjugated Increased (Investigations) | 3 | 3
Eosinophil Percentage Decreased (Investigations) | 3 | 0
Monocyte Count Increased (Investigations) | 3 | 0
Monocyte Percentage Decreased (Investigations) | 3 | 0
Protein Total Decreased (Investigations) | 3 | 0
Bacterial Test Positive (Investigations) | 2 | 1
Blood Alkaline Phosphatase Increased (Investigations) | 2 | 3
Blood Lactate Dehydrogenase Increased (Investigations) | 2 | 1
Blood Urine Present (Investigations) | 2 | 1
Electrocardiogram T Wave Abnormal (Investigations) | 2 | 0
Eosinophil Count Decreased (Investigations) | 2 | 0
Lymphocyte Percentage Decreased (Investigations) | 2 | 0
Plateletcrit Decreased (Investigations) | 2 | 0
Red Blood Cells Urine Positive (Investigations) | 2 | 4
Alanine Aminotransferase Abnormal (Investigations) | 1 | 1
Alpha Hydroxybutyrate Dehydrogenase Increased (Investigations) | 1 | 0
Basophil Count Increased (Investigations) | 1 | 0
Basophil Percentage Increased (Investigations) | 1 | 0
Blood Chloride Decreased (Investigations) | 1 | 0
Blood Cholinesterase Decreased (Investigations) | 1 | 0
Blood Creatine Phosphokinase Increased (Investigations) | 1 | 0
Blood Creatinine Increased (Investigations) | 1 | 2
Blood Pressure Systolic Decreased (Investigations) | 1 | 0
Blood Pressure Systolic Increased (Investigations) | 1 | 0
Blood Sodium Decreased (Investigations) | 1 | 0
Breath Sounds Abnormal (Investigations) | 1 | 0
Electrocardiogram St-T Segment Abnormal (Investigations) | 1 | 0
Fibrin D Dimer Increased (Investigations) | 1 | 1
Heart Rate Decreased (Investigations) | 1 | 0
Mean Cell Haemoglobin Increased (Investigations) | 1 | 0
Monocyte Count Decreased (Investigations) | 1 | 0
Mononuclear Cell Count Abnormal (Investigations) | 1 | 0
Platelet Distribution Width Decreased (Investigations) | 1 | 0
Prealbumin Decreased (Investigations) | 1 | 0
Protein Urine Present (Investigations) | 1 | 0
Prothrombin Level Decreased (Investigations) | 1 | 0
Prothrombin Time Ratio Decreased (Investigations) | 1 | 0
Sinus Rhythm (Investigations) | 1 | 0
Staphylococcus Test Positive (Investigations) | 1 | 0
Weight Decreased (Investigations) | 1 | 1
White Blood Cells Urine Positive (Investigations) | 1 | 3
Alpha 1 Foetoprotein Increased (Investigations) | 0 | 1
Aspartate Aminotransferase Abnormal (Investigations) | 0 | 1
Bilirubin Conjugated Abnormal (Investigations) | 0 | 1
Blood Albumin Abnormal (Investigations) | 0 | 1
Blood Bilirubin Abnormal (Investigations) | 0 | 2
Blood Potassium Increased (Investigations) | 0 | 1
Body Temperature Increased (Investigations) | 0 | 1
Crystal Urine Present (Investigations) | 0 | 1
Ejection Fraction Decreased (Investigations) | 0 | 1
Electrocardiogram Rr Interval Prolonged (Investigations) | 0 | 1
Electrocardiogram T Wave Amplitude Decreased (Investigations) | 0 | 1
Electrocardiogram T Wave Inversion (Investigations) | 0 | 1
Red Blood Cell Count Increased (Investigations) | 0 | 3
Total Bile Acids Increased (Investigations) | 0 | 1
Urinary Sediment Present (Investigations) | 0 | 1
Abdominal Pain Upper (Gastrointestinal disorders) | 39 | 39
Abdominal Pain (Gastrointestinal disorders) | 28 | 44
Nausea (Gastrointestinal disorders) | 20 | 12
Abdominal Distension (Gastrointestinal disorders) | 17 | 16
Constipation (Gastrointestinal disorders) | 17 | 18
Vomiting (Gastrointestinal disorders) | 9 | 8
Abdominal Tenderness (Gastrointestinal disorders) | 8 | 9
Mouth Ulceration (Gastrointestinal disorders) | 6 | 0
Aphthous Stomatitis (Gastrointestinal disorders) | 4 | 0
Ascites (Gastrointestinal disorders) | 4 | 4
Diarrhoea (Gastrointestinal disorders) | 4 | 4
Dyspepsia (Gastrointestinal disorders) | 4 | 4
Stomatitis (Gastrointestinal disorders) | 3 | 0
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 3 | 1
Dysphagia (Gastrointestinal disorders) | 2 | 0
Gastritis (Gastrointestinal disorders) | 2 | 1
Haemorrhoids (Gastrointestinal disorders) | 2 | 0
Abdominal Discomfort (Gastrointestinal disorders) | 1 | 0
Cheilitis (Gastrointestinal disorders) | 1 | 0
Dental Caries (Gastrointestinal disorders) | 1 | 0
Flatulence (Gastrointestinal disorders) | 1 | 2
Gastric Ulcer (Gastrointestinal disorders) | 1 | 1
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 1 | 3
Gingival Inflammation (Gastrointestinal disorders) | 1 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 1
Hyperchlorhydria (Gastrointestinal disorders) | 1 | 0
Intra-Abdominal Haemorrhage (Gastrointestinal disorders) | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 1 | 0
Oral Pain (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Peritoneal Haemorrhage (Gastrointestinal disorders) | 1 | 0
Proctalgia (Gastrointestinal disorders) | 1 | 0
Rectal Haemorrhage (Gastrointestinal disorders) | 1 | 0
Toothache (Gastrointestinal disorders) | 1 | 0
Varices Oesophageal (Gastrointestinal disorders) | 1 | 0
Anal Haemorrhage (Gastrointestinal disorders) | 0 | 1
Duodenal Perforation (Gastrointestinal disorders) | 0 | 1
Enterocolitis (Gastrointestinal disorders) | 0 | 1
Epigastric Discomfort (Gastrointestinal disorders) | 0 | 1
Eructation (Gastrointestinal disorders) | 0 | 1
Gingival Ulceration (Gastrointestinal disorders) | 0 | 1
Haematemesis (Gastrointestinal disorders) | 0 | 1
Intestinal Obstruction (Gastrointestinal disorders) | 0 | 1
Lower Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 1
Melaena (Gastrointestinal disorders) | 0 | 1
Pyrexia (General disorders) | 28 | 52
Puncture Site Pain (General disorders) | 14 | 14
Fatigue (General disorders) | 9 | 14
Chills (General disorders) | 4 | 2
Influenza Like Illness (General disorders) | 4 | 0
Non-Cardiac Chest Pain (General disorders) | 3 | 3
Oedema (General disorders) | 2 | 2
Oedema Peripheral (General disorders) | 2 | 2
Application Site Burn (General disorders) | 1 | 0
Asthenia (General disorders) | 1 | 1
Catheter Site Discolouration (General disorders) | 1 | 0
Chest Discomfort (General disorders) | 1 | 1
Effusion (General disorders) | 1 | 0
Impaired Healing (General disorders) | 1 | 0
Necrosis (General disorders) | 1 | 0
Pneumatosis (General disorders) | 1 | 0
Thirst (General disorders) | 1 | 0
Vessel Puncture Site Pain (General disorders) | 1 | 1
Feeling Cold (General disorders) | 0 | 1
Multi-Organ Failure (General disorders) | 0 | 1
Pneumonia (Infections and infestations) | 10 | 7
Urinary Tract Infection (Infections and infestations) | 10 | 7
Influenza (Infections and infestations) | 3 | 1
Nasopharyngitis (Infections and infestations) | 3 | 0
Sepsis (Infections and infestations) | 3 | 2
Upper Respiratory Tract Infection (Infections and infestations) | 3 | 3
Herpes Zoster (Infections and infestations) | 2 | 0
Liver Abscess (Infections and infestations) | 2 | 2
Wound Infection (Infections and infestations) | 2 | 0
Abdominal Infection (Infections and infestations) | 1 | 1
Body Tinea (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Diarrhoea Infectiouis (Infections and infestations) | 1 | 0
Ear Infection (Infections and infestations) | 1 | 0
Groin Abscess (Infections and infestations) | 1 | 0
Hepatic Infection (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 1 | 1
Lung Infection (Infections and infestations) | 1 | 0
Neutropenic Sepsis (Infections and infestations) | 1 | 0
Oral Candidiasis (Infections and infestations) | 1 | 0
Oral Herpes (Infections and infestations) | 1 | 0
Otitis Media (Infections and infestations) | 1 | 0
Post Procedural Infection (Infections and infestations) | 1 | 0
Pulmonary Tuberculosis (Infections and infestations) | 1 | 0
Septic Shock (Infections and infestations) | 1 | 1
Sinusitis (Infections and infestations) | 1 | 0
Subcutaneous Abscess (Infections and infestations) | 1 | 0
Tonsillitis (Infections and infestations) | 1 | 0
Tooth Infection (Infections and infestations) | 1 | 0
Urosepsis (Infections and infestations) | 1 | 0
Bacterial Infection (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 0 | 2
Febrile Infection (Infections and infestations) | 0 | 1
Folliculitis (Infections and infestations) | 0 | 1
Injection Site Abscess (Infections and infestations) | 0 | 1
Paronychia (Infections and infestations) | 0 | 1
Peritonitis (Infections and infestations) | 0 | 1
Pyelonephritis Acute (Infections and infestations) | 0 | 1
Rhinitis (Infections and infestations) | 0 | 1
Viral Infection (Infections and infestations) | 0 | 1
Procedural Pain (Injury, poisoning and procedural complications) | 22 | 28
Wound Complication (Injury, poisoning and procedural complications) | 6 | 4
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Muscle Strain (Injury, poisoning and procedural complications) | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 1 | 0
Post Procedural Complication (Injury, poisoning and procedural complications) | 1 | 2
Post Procedural Discharge (Injury, poisoning and procedural complications) | 1 | 1
Postoperative Wound Complication (Injury, poisoning and procedural complications) | 1 | 2
Procedural Intestinal Perforation (Injury, poisoning and procedural complications) | 1 | 0
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 1 | 0
Thermal Burn (Injury, poisoning and procedural complications) | 1 | 0
Brachial Plexus Injury (Injury, poisoning and procedural complications) | 0 | 1
Foreign Body (Injury, poisoning and procedural complications) | 0 | 1
Post Procedural Haematoma (Injury, poisoning and procedural complications) | 0 | 2
Post Procedural Inflammation (Injury, poisoning and procedural complications) | 0 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 17 | 12
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 13
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 4
Hiccups (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary Haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory Tract Irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypopneoa (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Oropharyngeal Plaque (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Decreased Appetite (Metabolism and nutrition disorders) | 19 | 11
Hypokalaemia (Metabolism and nutrition disorders) | 6 | 11
Hypoalbuminaemia (Metabolism and nutrition disorders) | 5 | 6
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 3 | 0
Gout (Metabolism and nutrition disorders) | 1 | 1
Hypercarotinaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 5
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 1
Hypochloraemia (Metabolism and nutrition disorders) | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1
Hypertension (Vascular disorders) | 15 | 16
Hypotension (Vascular disorders) | 3 | 3
Haematoma (Vascular disorders) | 2 | 1
Embolism Venous (Vascular disorders) | 1 | 0
Flushing (Vascular disorders) | 1 | 0
Haemorrhage (Vascular disorders) | 1 | 0
Vasculitis (Vascular disorders) | 1 | 0
Phlebitis (Vascular disorders) | 0 | 1
Liver Injury (Hepatobiliary disorders) | 6 | 3
Hepatic Function Abnormal (Hepatobiliary disorders) | 5 | 6
Portal Vein Thrombosis (Hepatobiliary disorders) | 3 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 2 | 4
Biliary Dilatation (Hepatobiliary disorders) | 1 | 0
Cholecystitis Acute (Hepatobiliary disorders) | 1 | 1
Hepatic Cirrhosis (Hepatobiliary disorders) | 1 | 1
Hepatic Failure (Hepatobiliary disorders) | 1 | 0
Hepatic Infarction (Hepatobiliary disorders) | 1 | 0
Hepatic Pain (Hepatobiliary disorders) | 1 | 3
Bile Duct Obstruction (Hepatobiliary disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Gallbladder Disorder (Hepatobiliary disorders) | 0 | 1
Hepatitis Toxic (Hepatobiliary disorders) | 0 | 1
Ischaemic Hepatitis (Hepatobiliary disorders) | 0 | 1
Jaundice (Hepatobiliary disorders) | 0 | 1
Portal Hypertension (Hepatobiliary disorders) | 0 | 1
Headache (Nervous system disorders) | 7 | 5
Dizziness (Nervous system disorders) | 4 | 1
Hepatic Encephalopathy (Nervous system disorders) | 3 | 1
Dysgeusia (Nervous system disorders) | 2 | 0
Cerebrovascular Accident (Nervous system disorders) | 1 | 1
Poor Quality Sleep (Nervous system disorders) | 0 | 1
Tremor (Nervous system disorders) | 0 | 2
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 4 | 6
Back Pain (Musculoskeletal and connective tissue disorders) | 3 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Flank Pain (Musculoskeletal and connective tissue disorders) | 2 | 2
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Rotator Cuff Syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Trigger Finger (Musculoskeletal and connective tissue disorders) | 1 | 0
Fistula (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1
Sinus Tachycardia (Cardiac disorders) | 3 | 0
Tachycardia (Cardiac disorders) | 3 | 2
Acute Myocardial Infarction (Cardiac disorders) | 2 | 0
Aortic Valve Incompetence (Cardiac disorders) | 1 | 0
Bundle Branch Block Right (Cardiac disorders) | 1 | 0
Cyanosis (Cardiac disorders) | 1 | 0
Left Ventricular Dysfunction (Cardiac disorders) | 1 | 0
Supraventricular Extrasystoles (Cardiac disorders) | 1 | 0
Angina Pectoris (Cardiac disorders) | 0 | 1
Atrial Fibrillation (Cardiac disorders) | 0 | 3
Atrioventricular Block Complete (Cardiac disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 5
Cardiac Ventricular Disorder (Cardiac disorders) | 0 | 1
Left Ventricular Hypertrophy (Cardiac disorders) | 0 | 1
Palpitations (Cardiac disorders) | 0 | 1
Urinary Retention (Renal and urinary disorders) | 2 | 1
Acquired Cystic Kidney Disease (Renal and urinary disorders) | 1 | 0
Chromaturia (Renal and urinary disorders) | 1 | 0
Dysuria (Renal and urinary disorders) | 1 | 3
Renal Disorder (Renal and urinary disorders) | 1 | 0
Renal Failure Acute (Renal and urinary disorders) | 1 | 2
Urinary Incontinence (Renal and urinary disorders) | 1 | 0
Diabetic Nephropathy (Renal and urinary disorders) | 0 | 1
Glomerulonephritis (Renal and urinary disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 4
Oliguria (Renal and urinary disorders) | 0 | 1
Proteinuria (Renal and urinary disorders) | 0 | 2
Pyuria (Renal and urinary disorders) | 0 | 1
Renal Impairment (Renal and urinary disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 6 | 5
Delirium (Psychiatric disorders) | 1 | 1
Depression (Psychiatric disorders) | 0 | 1
Addison's Disease (Endocrine disorders) | 1 | 0
Adrenocortical Insufficiency Acute (Endocrine disorders) | 1 | 0
Conjunctival Haemorrhage (Eye disorders) | 1 | 0
Vision Blurred (Eye disorders) | 1 | 0
Cataract (Eye disorders) | 0 | 1
Ocular Icterus (Eye disorders) | 0 | 1
Retinal Degeneration (Eye disorders) | 0 | 1
Drug Hypersensitivity (Immune system disorders) | 1 | 0
Immunosuppression (Immune system disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 0 | 1
Non-Small Cell Lung Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Infected Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tumour Haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI shall seek the Sponsor's prior review of publications, not before the multi-center publication has been published with Sponsor or 1 year from the date of Study completion/termination and only after review and comment by Sponsor. Proposed publication must be provided to Sponsor at least 60 days prior to submission to publisher. On Sponsor request, PI shall withhold a Publication from submission an additional 60 days to allow for the filing of a patent or any other protective actions available.

DOCUMENTS (2):
  • Study Protocol (2014-03-14): https://cdn.clinicaltrials.gov/large-docs/56/NCT02112656/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-16): https://cdn.clinicaltrials.gov/large-docs/56/NCT02112656/SAP_001.pdf